CLINICAL TRIAL: NCT00625651
Title: A Phase 1b/2 Study of AMG 655 in Combination With Modified FOLFOX6 and Bevacizumab for the First-Line Treatment of Subjects With Metastatic Colorectal Cancer
Brief Title: Phase 1b/2 Study of AMG 655 With mFOLFOX6 and Bevacizumab for First-Line Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20060464
Record Dates: First submitted 2008-02-14; First posted 2008-02-28 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-03

CONDITIONS: Metastatic Colorectal Cancer; Colon Cancer; Colorectal Cancer; Rectal Cancer
Keywords: Colon Cancer; Colorectal Cancer; Rectal Cancer; AMG 655; Bevacizumab; Modified FOLFOX6; mFOLFOX6; FOLFOX
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — conatumumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- AMG 655 Low Dose (Experimental): AMG 655 (low dose) + mFOLFOX6 + Bevacizumab
  Interventions: Drug: AMG 655; Drug: Modified FOLFOX6; Drug: Bevacizumab
- Placebo (Placebo Comparator): Placebo + mFOLFOX6 + Bevacizumab
  Interventions: Drug: Placebo; Drug: Modified FOLFOX6; Drug: Bevacizumab
- AMG 655 High Dose (Experimental): AMG 655 (high dose) + mFOLFOX6 + Bevacizumab
  Interventions: Drug: AMG 655; Drug: Modified FOLFOX6; Drug: Bevacizumab

INTERVENTIONS:
Drug: Placebo — Inactive dummy AMG 655 (to maintain blind)
  Arms: Placebo
Drug: AMG 655 — AMG 655 is an investigational, fully human monoclonal agonist antibody that selectively binds to Death Receptor-5 (DR5).
  Arms: AMG 655 High Dose; AMG 655 Low Dose
Drug: Modified FOLFOX6 — Combination treatment comprising oxaliplatin (85 mg/m2), leucovorin (400 mg/m2) and bolus 5-FU (400 mg/m2) and continuous IV 5-FU (2400 mg/m2)] administered by intravenous infusion once every 14 days (+3 days)
  Other Names: mFOLFOX6
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 5 mg/kg by intravenous infusion on day 1 of each 14 day cycle (+3 days).

SUMMARY:
This phase 1/2, multi-center, randomized, double-blind, placebo-controlled trial is designed to evaluate the efficacy and safety of AMG 655 when combined with mFOLFOX6 and bevacizumab compared with mFOLFOX6 and bevacizumab alone in subjects with previously untreated metastatic colorectal cancer (CRC).

The clinical benefit of AMG 655 in combination with mFOLFOX6 and bevacizumab will be measured by progression-free survival, objective response rate, time to response, duration of response, and overall survival. This study is also designed to evaluate the safety and tolerability of AMG 655 in combination with mFOLFOX6 and bevacizumab and to evaluate anti-AMG 655 antibody formation and the pharmacokinetics of AMG 655.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic adenocarcinoma of the colon or rectum.
* Subjects with measurable or unmeasurable disease
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Men or women at least 18 years of age
* Adequate hematologic, renal, hepatic and coagulation function

Exclusion Criteria:

* History or known presence of central nervous system (CNS) metastases
* Prior chemotherapy or other systemic therapy for advanced or metastatic CRC
* Any investigational agent or therapy for advanced or metastatic CRC
* Clinically significant cardiac disease
* Clinically significant peripheral neuropathy
* Active inflammatory bowel disease
* Recent gastrointestinal ulcer or hemorrhage
* Recent arterial thrombotic event or pulmonary embolus
* Recent history of clinically significant bleeding, bleeding diathesis, or coagulopathy
* Recent major surgical procedure or not yet recovered from major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Length of study

SECONDARY OUTCOMES:
Objective response rate | Length of study
Duration of response | Length of study
Time-to-response | Length of study
Overall survival | Length of study
AMG 655 pharmacokinetic parameters | Length of study
The incidence of anti-AMG 655 antibody formation | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (59):
- United States (59):
  - Research Site, Hot Springs, Arkansas
  - Research Site, Downey, California
  - Research Site, La Jolla, California
  - Research Site, Loma Linda, California
  - Research Site, Orange, California
  - Research Site, Rancho Mirage, California
  - Research Site, San Diego, California
  - Research Site, Denver, Colorado
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Harvey, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Great Falls, Montana
  - Research Site, Long Branch, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, Hudson, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Burlington, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Middletown, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pottsville, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Richardson, Texas
  - Research Site, Tyler, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Ogden, Utah
  - Research Site, Fairfax, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Vancouver, Washington

REFERENCES:
- [Background] Fuchs CS, Fakih M, Schwartzberg L, Cohn AL, Yee L, Dreisbach L, Kozloff MF, Hei YJ, Galimi F, Pan Y, Haddad V, Hsu CP, Sabin A, Saltz L. TRAIL receptor agonist conatumumab with modified FOLFOX6 plus bevacizumab for first-line treatment of metastatic colorectal cancer: A randomized phase 1b/2 trial. Cancer. 2013 Dec 15;119(24):4290-8. doi: 10.1002/cncr.28353. Epub 2013 Oct 1. PMID 24122767
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com